CLINICAL TRIAL: NCT07293533
Title: Estratificação de Risco em Cirurgia de revascularização miocárdica no Brasil: CABG - BraSCORE (Brazilian System for Cardiac Operative Risk Evaluation)
Brief Title: Brazilian System for Cardiac Operative Risk Evaluation CABG
Acronym: BRASCORE CABG
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Instituto Nacional de Cardiologia de Laranjeiras (Other); Beneficência Portuguesa de São Paulo (Other); Santa Casa de Misericórdia de Marília (Unknown); Professor Fernando Figueira Integral Medicine Institute (Other); Hospital do Coração de Messejana Dr. Carlos Alberto Studart (Unknown); Instituto de Cardiologia do Rio Grande do Sul (Other); Irmandade da Santa Casa de Misericordia de Curitiba (Other); Hospital Universitário do Maranhão - MA (Unknown); Hospital do Coração Alagoano Prof. Adib Jatene (Unknown); Irmandade da Santa Casa de Misericordia de Sao Paulo (Other); Hospital São Francisco de Assis na Providência de Deus - RJ (Unknown); Hospital Universitario Pedro Ernesto (Other); Cardiac Emergency Hospital of Pernambuco (Unknown); Hospital Geral de Cuiabá (Unknown); Hospital Beneficente Portuguesa de Belém (Unknown); Pronto-Socorro Cardiológico Universitário de Pernambuco (Unknown); Hospital Alberto Urquiza Wanderley de João Pessoa (Unknown); Hospital e Maternidade Marieta Konder Bornhausen (Unknown); Hospital Arquidiocesano Consul Carlos Renaux (Unknown); Hospital Universitário São Francisco na Providência de Deus (HUSF) (Unknown); Hospital Regional de Jundiaí (Unknown); Hospital Ruy Azeredo (Unknown); Hospital de Base São José do Rio Preto (Unknown); Hospital São Vicente de Paulo (Unknown); Hospital das Clínicas da UFMG (Unknown); Hospital de Cirurgia (Unknown); Hospital Universitário (USP Riberão Preto) (Unknown); Fundação Hospital do Coração Francisca Mendes (Unknown); Hospital Dom Helder Câmara (Unknown); Hospital Santa Casa de Curitiba (Unknown); Hospital São Vicente de Paulo - Jundiai (Unknown)
Responsible Party: Principal Investigator, Omar Asdrúbal Vilca Mejia, MD PhD, University of Sao Paulo General Hospital
Other Study IDs: 76508623.2.1001.0068; 7.933.450 (Registry Identifier: Ethical approval)
Record Dates: First submitted 2025-11-25; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: CABG-patients
Keywords: Databases; Database Management Systems; Coronary Artery Bypass; Predictions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Grouping relevant demographic and clinical information at specific stratified levels, and in correlation with the required resource sets, represents the possibility to adapt, improve, and innovate in cardiac surgery programs. In this path, the pursuit of implementing large databases for continuous improvement cycles becomes the foundation of the entire process. In Brazil, where structural and socioeconomic differences are significant, the standardization and sustainability of a large database become a major challenge. Projects like REPLICCAR (São Paulo Cardiovascular Surgery Registry) and BYPASS Registry, which were created to identify improvement opportunities, were temporary. The absence of a continuous multicenter registry makes it difficult to understand risk-adjusted patient outcomes and to implement cost-effective quality initiatives. For example, in 2022, the Ministry of Health launched the QualiSUS Cardio program, which began to consider hospital reimbursement not only in terms of surgical volume but also in relation to mortality, length of stay, and readmission rates after cardiac surgery. Changes like this already occur in various scenarios where payers, whether public or private, seek reimbursement through value-based models. However, for this to happen, the results need to be adjusted to patient risk. Otherwise, hospitals treating more severe patients would be at a disadvantage. This study aims to develop CABG-BraSCORE, a risk score to stratify patients referred for CABG surgery, adjusting outcomes to patient risk, and seeking continuous improvement for cardiac surgery programs in Brazil.

DETAILED DESCRIPTION:
Study Procedure: Data collection will be conducted from patient records, including demographic characteristics, preoperative status, surgical and postoperative data of CABG surgery, and follow-up up to 30 days post-discharge.

Centers with prospective data collection: Participants will be contacted 30 days after surgery and invited to participate in the study. The Free and Informed Consent Form (FICF) will be applied via telephone (Appendix 1). All FICF sessions will be recorded, downloaded, and stored according to the established study protocols.

Centers with retrospective data collection: Thirty days after surgery, it should be recorded whether there was a return visit to the outpatient clinic, readmission to the institution, the reason for readmission, such as surgical complications, stroke, surgical wound infection, myocardial infarction, and mortality at 30 days. All records should be consulted in the patient's medical record. If there is no information recorded about the patient's return visit, loss to follow-up should be considered. A loss of 20% was considered for the sample composition.

After the telephone FICF, a questionnaire (Appendix 2, within the Cardux platform's "Post-discharge Events" section) will be applied to gather information regarding readmissions, death, adverse events, among others, within 30 days after hospital discharge.

Patient data will be entered into the Cardux platform according to study protocol variables.

All inclusion steps will be guided by the coordinating center, providing clarification about the study protocol and ensuring its compliance, respecting the ethical and legal principles of the study.

* Risks to Participants Participants will be exposed to minimal risk as this study will not involve interventions, only a single telephone interview. Therefore, no risks to participants are anticipated, as the data collection will be entirely retrospective and the consent forms will be stored confidentially.
* Benefits to Participants: Participants will not receive any direct benefit from participating in this study. However, in the future, they might benefit from improved risk stratification for CABG surgeries, contributing to enhanced patient care and resource allocation.
* Cardux Platform Cardux platform will be used for data management and analysis. This platform facilitates real-time monitoring and auditing of data, ensuring consistency and accuracy. The platform also supports predictive modeling and quality assessment.
* Quality Audit of Records: To ensure data quality, a series of audits will be conducted. These audits will involve checking data completeness, consistency, and accuracy. Discrepancies will be resolved through communication with the participating centers.
* Data analysis will include statistical methods to evaluate risk factors and develop the BraSCORE. The model's performance will be validated and compared with existing international risk scores (EuroSCORE III and STS)
* Development of Machine Learning Algorithms Machine learning algorithms will be employed to develop predictive models for hospital mortality, readmission risk, and prolonged hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to isolated coronary artery bypass grafting at participating centers

Exclusion Criteria:

* Emergency or salvage CABG procedures.
* Associated procedures (e.g., valve surgery, aortic surgery).
* Missing mandatory data in the registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all consecutive patients undergoing isolated CABG at the participating centers during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | up to 3 months during hospital admission for CABG
  death occurring at any point during the hospitalization for surgery, even if after 30 days
30-day mortality | 30-days of the procedure
  death occurring after discharge from the hospital, but within 30-days of the procedure

SECONDARY OUTCOMES:
Prolonged Hospital Stay | postoperative hospital stay longer than 14 days
  Postoperative hospital stay longer than 14 days, excluding in-hospital deaths
30-day readmission | 30-days after surgery
  any unplanned admission for any reason within 30-days of CABG surgery discharge

OTHER OUTCOMES:
Data quality score | Assessment will be performed on registries that have completed a 30-day active data collection period.
  Data quality will be assessed using a composite Aggregate Data Quality Score (ADQ), calculated as the average of three metrics: 1) Completeness (>70% threshold): the percentage of mandatory fields populated, calculated as (Total non-missing values / Total possible values); 2) Consistency (>90% threshold): the percentage of fields free from logical contradictions (ex.: discharge before admission) and format errors; and 3) Accuracy (>90% threshold): the percentage of fields correctly reflecting the source electronic health record, as verified by periodic in-loco audit. The ADQ provides a single summary measure of overall registry data reliability.

CONTACTS AND LOCATIONS:
Overall Officials: BIANCA MARIA MAGLIA ORLANDI, Post doctoral resercher, Study Director
Locations (5):
- Brazil (5):
  - Hospital de Messejana, Fortaleza, Ceará
  - Hospital Alberto Urquiza Wanderley, João Pessoa, Paraíba
  - USP Heart Institute, São Paulo, São Paulo
  - Instituto Nacional de Cardiologia de Laranjeiras, Rio de Janeiro
  - Beneficência Portuguesa de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided
The Individual Participant Data (IPD) that support the findings of this study are not publicly available due to ethical restrictions imposed by the participating centers and the overseeing ethics committee (Comissão de Ética para Análise de Projetos de Pesquisa - CAPPesq). However, de-identified data may be made available to qualified researchers upon reasonable request, subject to approval by CAPPesq and the execution of a data sharing agreement.

REFERENCES:
- [Background] Atik FA. Registries and Evidence-Based Medicine. Arq Bras Cardiol. 2024 Aug 2;121(6):e20240330. doi: 10.36660/abc.20240330. eCollection 2024. No abstract available. English, Portuguese. PMID 39109690
- See also: Study website — https://www.cardux.net/brascore